CLINICAL TRIAL: NCT02048072
Title: Funktionelle Evaluation Des Autonomen Nervensystems im Zusammenhang Mit Der Erstmaligen Einnahme Von 0,5mg Fingolimod (Gilenya) Bei Patienten Mit schubförmig Verlaufender Multipler Sklerose
Brief Title: Evaluation of the Autonomic Nervous System During First-dosing With 0.5mg of Fingolimod (Gilenya) in Patients With Relapsing-remitting MS
Acronym: ANSG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jochen Vehoff (Other)
Responsible Party: Sponsor-Investigator, Jochen Vehoff, Dr. med. Jochen Vehoff, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANSG 1.8
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis; Autonomic Nervous System Dysfunction
Keywords: relapsing remitting; multiple sclerosis; fingolimod; Gilenya; autonomic nervous system
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gilenya (Experimental): Autonomic testing during first dose adminstration of Gilenya.
  Interventions: Drug: Gilenya

INTERVENTIONS:
Drug: Gilenya — Autonomic testing during first dose administration of Gilenya.

SUMMARY:
This study is designed to primarily evaluate the impact of Gilenya (Fingolimod) on the autonomic nervous system in patients being treated for the first time with Gilenya (Fingolimod). Effects on the cardiovascular system will be studied as well. The study is conducted to answer the question, if, and if yes, what impact the treatment with Gilenya (Fingolimod) has on the autonomic nervous system. To our knowledge little is known about the effects of Gilenya (Fingolimod) on the autonomic nervous system. We do know of rare, but potentially clinically and therapeutically relevant cardiovascular adverse events of Gilenya (Fingolimod). From a scientific point of view the mechanisms by which this is mediated are of interest. Maybe a better understanding of these mechanisms might even be of clinical relevance (e.g. risk stratification).

The impact of Gilenya (Fingolimod) on the autonomic nervous system is quantitavely measured, using a state-of-the-art technique. Non-invasive blood pressure measurement is performed with the Finometer Pro (Finapres Medical Systems, NL) under different paradigms (breathing at rest, deep breath, valsalva maneuver, active standing). In addition the sympathetic skin reaction is performed. The non-invasive blood pressure measurements are done by continuous, plethysmographic blood pressure measurement at the index finger, while the patient is performing the tasks mentioned above. By interpreting the blood pressure curve, heart rate and blood pressure variability are calculated. The sympathetic skin reaction consists of measuring the change of electric conductibility of the skin (palms and soles) after an electric stimulus of a peripheral nerve. These parameters allow to assess the functionality of four important autonomic functional systems (orthostasis, sympathetic adrenergic, sympathetic cholinergic, parasympathetic cholinergic). Normative data has been acquired in our lab.

Our hypothethis is, that there will be a change of heart rate variability at t4,5h compared to baseline (t0) for the parameter "RMSSD" under "normal breathing".

ELIGIBILITY:
Inclusion Criteria:

* indication for treatment with Gilenya according label
* treatment with Gilenya intended
* no contraindications for the treatment with Gilanya
* all safety-aspects have been fullfilled
* age between 18 and 60 years
* written consent is given

Exclusion Criteria:

* relapse during the last 30 days befor randomization
* steroids within 30 days before randomization
* heart rhythm disturbance
* new or currently changed dose (last 4 weeks) of bata-blockers, calcium antagonists, antidepressants or antiarrhythmics
* diabetes mellitus
* polyneuropathy
* missing consent
* pregnancy
* lactation period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Vehoff, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 21.08.2013 Last patient out: 16.06.2015
Groups:
- Gilenya: Gilenya 0.5mg p.o. once daily
Period: Overall Study
Arm/Group | Gilenya
Started | 33
Completed | 29
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gilenya
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.57 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 8
Region of Enrollment [Number; unit: participants]
  Switzerland | 33
EDSS [Mean (Standard Deviation); unit: units on a scale] — Expanded Disability Status Scale Range 0-10 (no disability - death due to Multiple Sclerosis)
  units on a scale | 1.75 (1.16)
Weight [Mean (Standard Deviation); unit: kg] | 71.18 (13.18)
Height [Mean (Standard Deviation); unit: cm] | 168.72 (7.98)
Body temperature [Mean (Standard Deviation); unit: °C] | 36.58 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: RMSSD Normal Breathing
Description: Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR or pulse intervals.
  It is calculated as the square root of the mean of the squares of the successive differences between adjacent RR intervals or pulse intervals.
  In this study pulse intervals were measured non-invasively during five minutes, while subjects were supine, breathing regularly.
  Measurements were done at two timepoints t=0 and t=4,5hours. RMSSD was compared between these two timepoints.
Time Frame: t-4,5 hours
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Gilenya
Number analyzed (Participants) | 32
milliseconds | 14.10 [2.56 to 25.65]
Statistical Analysis 1: Comparison: Gilenya; Test type: Superiority or Other; p = 0.02, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Gilenya
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 1/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilenya (N=33)
AV-Block Mobitz II / AV-Block III° (Cardiac disorders) | 1 (1)
worsening of neuropsychological symptoms (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilenya (N=33)
exacerbation of migraines (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No